CLINICAL TRIAL: NCT05610553
Title: Application of 3D Printing Guide Plate in Percutaneous Disc Decompression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TTK03
Record Dates: First submitted 2022-10-30; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-09

CONDITIONS: Lumbar Disc Herniation; Radiculopathy; Percutaneous Disc Decompression; 3D Printing Guide Plate; Radicular Pain; Low Back Pain; Discogenic Pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy; Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printing guide plate group (Experimental): 3D-printed customized guide plate will be used to guide the puncture in percutaneous disc decompression surgeries.
  Interventions: Other: 3D printing guide plate
- Conventional guidance group (Active Comparator): The surgeons would place the needle according to his/her previous experience under the guidance of C-arm fluoroscopy or CT.
  Interventions: Other: Conventional guidance

INTERVENTIONS:
Other: 3D printing guide plate — 3D-printed customized guide plate will be used to guide the puncture in percutaneous disc decompression surgeries to help to reduce intra-operative radiation, puncture time, etc..
  Arms: 3D printing guide plate group
Other: Conventional guidance — The surgeons would place the needle according to his/her previous experience under the guidance of C-arm fluoroscopy or CT.
  Arms: Conventional guidance group

SUMMARY:
Application of 3D printing guide plate in percutaneous disc decompression

DETAILED DESCRIPTION:
This study applies 3D-printed customized guide plate in assisting the accurate puncture in percutaneous disc decompression, in patients with low back pain, lumbosacral radicular pain, disogenic pain, lumbar disc herniation, disc degeneration, etc. This technique can shorten reduce the intra-operative radiation, and do not affect the surgical outcome.

This study involved diseases such as lumbar disc herniation (LDH), disc degeneration, etc. Percutaneous disc decompression surgeries are effective treatments for these disease. Needle Puncture is the key technology in percutaneous disc decompression surgeries.

In the past when there were no customized guides, the surgeons would place the needle according to his/her previous experience under the guidance of C-arm fluoroscopy or CT. If the position of the needles is not satisfactory, repeated procedure will be performed. This would lead to an increase in the duration of surgery and intra-operative radiation, which is detrimental to both the surgeon and the patient. This problem could be well solved by applying the 3D printing guide plate.

The key processes for the 3D printing guide plate procedure: the model of the spine or bone is established according to the patient's CT scan data to prepare the customized guide plate, then sterilize them for future use. The final position of needle is confirmed by C-arm fluoroscopy or CT or evoked pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Pain lasting ≥12 weeks;
3. The previous failure of conservative management such as physiotherapy, exercise therapy, or analgesic medications;
4. Pain intensity≥4 out of 10 on the numerical rating scale (NRS);
5. Availability of computed tomography/magnetic resonance imaging findings of pathology concordant with the side and level of their clinical features;
6. Agree with percutaneous disc decompression.

Exclusion Criteria:

1. Patient refusal to participate in the study;
2. Pregnant or nursing;
3. Allergies to local anesthetics, contrast dyes or steroids;
4. Significant anatomic deformity (either congenital or acquired) making it difficult to access the target as evidenced by computed tomography/magnetic resonance imaging;
5. Patients with platelet dysfunction, bleeding disorder or continuing anticoagulant treatment;
6. Systemic infection;
7. Injection site infection;
8. Unstable medical or psychiatric condition;
9. Unable to tolerate the surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-12-10 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
C-arm fluoroscopy times | Intraoperative
  Numbers of using C-arm fluoroscopy

SECONDARY OUTCOMES:
Puncture time | Intraoperative
  Time from the first puncture to the last puncture
Numerical rating scale (NRS) | Postoperative 1 day, 2 weeks, 1 month
  NRS at 1 day, 2 weeks, 1 month after the operation
MacNab | Postoperative 1 months
  Patient satisfaction using the modified MacNab criteria
Complications | Intraoperative
  Complication like nerve injury, blood, hemotoma, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Pain medicine center of Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No